CLINICAL TRIAL: NCT06710353
Title: The Effect of Preoperative Albumin Administration on Postoperative Acute Kidney Injury in Pediatric Patients With Hypoalbuminemia Undergoing Cardiac Surgery: A Prospective Randomized Clinical Trial
Brief Title: The Effect of Preoperative Albumin Administration on Postoperative Acute Kidney Injury in Pediatric Patients With Hypoalbuminemia Undergoing Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ji-Hyun Lee, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H2410-094-1578
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Acute Kidney Injury; Pediatric Cardiac Surgery
MeSH Terms: conditions — Acute Kidney Injury | interventions — Crystalloid Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Albumin group (Experimental): A 20% albumin solution is administered over a period of one hour, starting at the time of anesthesia induction.
- Control group (Placebo Comparator): The same volume of crystalloid solution as the administered albumin is infused.

INTERVENTIONS:
Drug: Albumin solution — A 20% albumin solution is administered over one hour starting from the induction of anesthesia, using the following formula:
  (4.0-preoperative serum albumin (g/dL))×plasma volume (kg×0.65-0.8 dL)
Drug: Crystalloid solutions — The same volume of crystalloid solution as the administered albumin is infused.

SUMMARY:
The study aims to evaluate whether preoperative albumin supplementation in pediatric patients with hypoalbuminemia undergoing cardiac surgery can reduce inflammatory responses and prevent acute kidney injury (AKI) following cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients under 7 years of age undergoing cardiac surgery with cardiopulmonary bypass
* Preoperative serum albumin level of 4.0 g/dL or lower

Exclusion Criteria:

* abnormal preoperative creatinine level
* history of dialysis
* liver dysfunction
* diabetes
* history of hypersensitivity to albumin
* coagulation disorders

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 190 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of acute kidney injury (AKI) | assessed up to postoperative day 7
  The difference in the incidence of acute kidney injury (AKI) between groups, as measured by the KDIGO criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided